CLINICAL TRIAL: NCT04862832
Title: Reduction of Thermal Pain From a Personalized Musical Intervention : Effect of Musical Preference
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association de Musicothérapie Applications et Recherches Cliniques (Other)
Collaborators: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MUSEC
Record Dates: First submitted 2021-04-16; First posted 2021-04-28 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Pain
Keywords: Pain; Anxiety; Musical intervention; Web app-based
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPT - LLM - MLM (Experimental): On day 1: CPT On day 2: LLM On day 3: MLM
  Interventions: Other: Music intervention
- CPT - MLM - LLM (Experimental): On day 1: CPT On day 2: MLM On day 3: LLM
  Interventions: Other: Music intervention

INTERVENTIONS:
Other: Music intervention — The cold pressor test will consist in the immersion of the participants' arm in 10 degrees circulating water for two minutes.
  The music sequences will be all 20 minutes, instrumental, professionally recorded in the studio and composed specifically for the Music Care application and are thus unfamiliar to participants. There will be two music conditions: the most-liked-music (MLM) and least-liked-music (LLM) conditions.
  Other Names: Cold Pressor Test (CPT)

SUMMARY:
This is a randomized, 3-days study with the objective to compare the modulation of pain from our musical intervention to the CPT-induced analgesia and silence. The mean pain felt before and after CPT, the silence, and at three times points for the music conditions, 2.20 minutes, 11.30 minutes and 20 minutes, will be evaluated.

Based on previous data, the sample size has been estimated, and 30 participants will be enrolled.

They will undergo four conditions: CPT, silence, Most-Liked Music (MLM) and Least-Liked Music.

The music used will be Music Care, a personalized musical intervention used in clinical settings. It has a U shape in six sections that each have different tempi, number of instruments and volume.

There will be two music conditions: the most-liked-music (MLM) and least-liked-music (LLM) conditions. The sequence rated the highest will be listened to during the MLM and the one rated the lowest will be listened during the LLM condition. MLM will be considered as a score between 7 and 10 on the preference scale. LLM will be considered as a score between 0 and 4.

The cold pressor test will consist in the immersion of the participants' arm in 10 degrees circulating water for two minutes.

The silence condition will consist of six minutes in which the participants stay seated on the examination chair without access to their phones or other provided distractions.

There will be three testing days for each participants. They will be seated in a comfortable chair in a quiet room. The first day, before the pain tests started, consent form will be read and signed by the participants. After, the MLM and LLM will be determined. Then, the sociodemographic questionnaire, the two State Trait Anxiety Inventory (STAI) subscales, Beck Depression Inventory (BDI) and Pain Catastrophizing Scale (PCS) will be administered. Finally, a first two minutes pain test will be performed (T1), the CPT and a second pain test (T2).

The second and third day will consist of first the STAI, the state subscale, the silence condition and then one music condition. The order of music condition will be randomized. The silence condition will consist of a first pain test (T3 or T8), six minutes of silence and then a second pain test (T4 or T9). Those 6 minutes will be chosen in order to equal the duration between the end of the first pain test and the start of the second one of the music intervention condition. In fact, for the music condition, whether it's the MLM or LLM, the first pain tests will be performed at 2.20 minutes after the music started (T5 or T10). The second will be after the relaxation phase at 11.30 minutes (T6 or T11) and the third after the whole 20-minutes cycle (T6 or T12). A post music condition score of the MLM and LLM on the same preference scale as the selection will be administered.

Quantitative data will be described using mean, standard deviation, median, extreme values (minimum and maximum) and the number of missing data.

Qualitative data will be described by their distributions in terms of numbers and percentages by class as well as the number of missing data.

The normality condition will be verified using the Shapiro-Wilk test. Quantitative variables will be compared by the paired Student test if conditions were checked or by the non-parametric test of the signed Wilcoxon ranks, as part of the comparison of 2 modalities. The quantitative variables will be compared between the 3 conditions using a repeated-measure ANOVA or Friedman test.

Tests will be bilateral, with a threshold of 5%.

DETAILED DESCRIPTION:
Background: Music is used as a management technique for pain in multiple clinical settings. Music-induced analgesia (MIA) seems to be using the endogenous descending pain modulatory system. This latter is demonstrated by the The Cold Pressor Test (CPT), used here alongside silence as a control condition for MIA.

Study design: This is a randomized, 3-days study with the objective to compare the modulation of pain from our musical intervention to the CPT-induced analgesia and silence.

Objectives: The objective of this study will be to compare the modulation of pain from our musical intervention to the CPT-induced analgesia and silence. In addition, the difference in pain modulation from the most-liked music and least-liked music conditions will be evaluated. It is predicted that most liked music will reduce pain perception in a similar fashion than the CPT and more than the least liked music and silence.

The mean pain felt before and after CPT, the silence, and at three times points for the music conditions, 2.20 minutes, 11.30 minutes and 20 minutes, will be compared.

Participants: Based on previous data, the sample size has been estimated, and 30 participants will be enrolled.

Intervention: Each participant will undergo four conditions: CPT, silence, Most-Liked Music (MLM) and Least-Liked Music.

The music used will be Music Care, a personalized musical intervention used in clinical settings. It has a U shape in six sections that each have different tempi, number of instruments and volume.

There will be two music conditions: the most-liked-music (MLM) and least-liked-music (LLM) conditions. The sequence rated the highest will be listened to during the MLM and the one rated the lowest will be listened during the LLM condition. MLM will be considered as a score between 7 and 10 on the preference scale. LLM will be considered as a score between 0 and 4.

The cold pressor test will consist in the immersion of the participants' arm in 10 degrees circulating water for two minutes.

The silence condition will consist of six minutes in which the participants stay seated on the examination chair without access to their phones or other provided distractions.

Measures: There will be three testing days for each participants. They will be seated in a comfortable chair in a quiet room. The first day, before the pain tests started, consent form will be read and signed by the participants. After, the MLM and LLM will be determined. Then, the sociodemographic questionnaire, the two STAI subscales, BDI and PCS will be administered. Finally, a first two minutes pain test will be performed (T1), the CPT and a second pain test (T2).

The second and third day will consist of first the STAI, the state subscale, the silence condition and then one music condition. The order of music condition will be randomized. The silence condition will consist of a first pain test (T3 or T8), six minutes of silence and then a second pain test (T4 or T9). Those 6 minutes will be chosen in order to equal the duration between the end of the first pain test and the start of the second one of the music intervention condition. In fact, for the music condition, whether it's the MLM or LLM, the first pain tests will be performed at 2.20 minutes after the music started (T5 or T10). The second will be after the relaxation phase at 11.30 minutes (T6 or T11) and the third after the whole 20-minutes cycle (T6 or T12). A post music condition score of the MLM and LLM on the same preference scale as the selection will be administered.

Statistical methods: Quantitative data will be described using mean, standard deviation, median, extreme values (minimum and maximum) and the number of missing data.

Qualitative data will be described by their distributions in terms of numbers and percentages by class as well as the number of missing data.

The normality condition will be verified using the Shapiro-Wilk test. Quantitative variables will be compared by the paired Student test if conditions were checked or by the non-parametric test of the signed Wilcoxon ranks, as part of the comparison of 2 modalities. The quantitative variables will be compared between the 3 conditions using a repeated-measure ANOVA or Friedman test.

Tests will be bilateral, with a threshold of 5%.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults

Exclusion Criteria:

* musicians with knowledge of music theory
* diagnosed and taking medication for chronic pain
* skin problems
* psychological or neurological pathologies

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Pain level change from baseline to the end of music intervention | Collected before the music starts (considered as baseline), and after the whole 20-minutes cycle.
  Pain level measured using a Computerized Visual Analogue Scale (VAS) from 0: "no pain" to 100: "most intense pain tolerable".

SECONDARY OUTCOMES:
Pain level change from baseline to the beginning of music intervention | Collected before the music starts (considered as baseline) and 2.20 minutes after the music start.
  Pain level measured using a Computerized Visual Analogue Scale (VAS) from 0: "no pain" to 100: "most intense pain tolerable".
Pain level change from baseline to the relaxation phase of music intervention | Collected before the music starts (considered as baseline) and after the relaxation phase at 11.30 minutes.
  Pain level measured using a Computerized Visual Analogue Scale (VAS) from 0: "no pain" to 100: "most intense pain tolerable".
Perception of time | 20 minutes after music starts
  Under both music conditions, the duration of the session will not be communicated to the participants. At the end of the musical intervention sequence, they will be asked how long it had lasted according to their opinion.

CONTACTS AND LOCATIONS:
Locations (1):
- Sherbrooke University Hospital Centre, Sherbrooke, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soyeux O, Marchand S. A web app-based music intervention reduces experimental thermal pain: A randomized trial on preferred versus least-liked music style. Front Pain Res (Lausanne). 2023 Jan 16;3:1055259. doi: 10.3389/fpain.2022.1055259. eCollection 2022. PMID 36726374